CLINICAL TRIAL: NCT02673112
Title: Study of an Exercise Program (STEP) for Youth With Concussion
Acronym: STEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Sara Chrisman, Assistant Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00000023
Record Dates: First submitted 2016-01-26; First posted 2016-02-03 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Persistent Concussion Symptoms
Keywords: Concussion; mild traumatic brain injury; post concussion syndrome; child
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- STEP-mhc + LS (Experimental): Subjects will be asked to perform exercise at 80% of the heart rate threshold determined using the Balke protocol for 5 minutes greater than their measured minutes of MVPA/day at baseline (Subthreshold exercise program). They will also be given a light stretching protocol (5 stretches). The exercise intervention will last for 6 weeks and will be supported by weekly health coaching.
  Interventions: Behavioral: Subthreshold exercise (STEP) with mobile health coaching; Behavioral: Light stretching (LS)
- LS alone (Active Comparator): Subjects will be given a light stretching program alone (5 stretches). The exercise program will last for 6 weeks.
  Interventions: Behavioral: Light stretching (LS)

INTERVENTIONS:
Behavioral: Subthreshold exercise (STEP) with mobile health coaching — Aerobic exercise program performed below the HR threshold that causes symptoms and administered by an RA using mobile health coaching
  Arms: STEP-mhc + LS
Behavioral: Light stretching (LS) — Brief daily stretching routine.

SUMMARY:
To compare the efficacy of a sub-threshold aerobic exercise intervention provided with mobile health coaching (STEP-mhc) and a light stretching program (LS) to LS alone for 11-18 yo youth with persistent concussion symptoms.

DETAILED DESCRIPTION:
This is a minimal risk randomized controlled trial whose aim is to test the efficacy of an exercise intervention (STEP) for youth 11-18 yo with persistent concussive symptoms (1-6 months inclusive). The investigators are utilizing an active control (light stretching). The primary outcome will be concussion symptoms measured with the Health-Behavior Inventory (HBI) in the first month after randomization. Long-term efficacy will be examined using standardized measures of quality of life and function over 6 months, and potential mediators will be explored including brain derived neurotrophic factor (BDNF), fear-avoidance and physical fitness. Physical activity will be measured with accelerometry to evaluate fidelity.

ELIGIBILITY:
Inclusion Criteria:

* Sports-related concussion that occurred 1-6 months inclusive prior to the start of the study, and was diagnosed by a clinician trained in concussion management consistent with the Zurich definition of concussion ("a complex pathophysiological process affecting the brain, induced by biomechanical forces [that] results in a graded set of clinical symptoms that may or may not involve loss of consciousness")
* Persistent symptoms as defined by the presence of at least 2 concussive symptoms (from the Health Behavior Inventory, or HBI) at the time of recruitment which were not present prior to injury
* 11 to 18 years of age (inclusive) at time of recruitment

Exclusion Criteria:

* Non-English speaking youth or parents
* Unwilling or unable to travel to Seattle Children's Hospital or Seattle Children's Research Institute twice during the course of the study
* Cervical spine or vestibular issues requiring further targeted intervention
* Other injuries or medical conditions in addition to concussion which would preclude vigorous exercise
* Psychiatric hospitalization in the year prior to enrollment
* Significant cognitive deficits such as mental retardation or autism
* Lack of worsening of concussive symptoms with exertion
* Significant abnormalities on routine brain imaging.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2016-04; Primary Completion 2017-09 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Health Behavior Inventory (HBI) | Baseline, Weekly from 1-6 weeks, 3 months, 6 months
  Measure change in concussion symptoms from the baseline evaluation to post-intervention (6 weeks) using HBI.

SECONDARY OUTCOMES:
PedsQL | Baseline, 6 weeks, 3 and 6 months
  Health related quality of life
Fear of Pain Questionniare (FOPQ), child and parent | Trajectory from baseline, 6 weeks, 3 months, 6 months
  Measure of fear avoidance
Moderate-vigorous physical activity (MVPA) | Baseline and 6 weeks
  Hip-mounted research grade accelerometry

CONTACTS AND LOCATIONS:
Overall Officials: Sara P Chrisman, MD MPH, Principal Investigator — Seattle Childrens Research Institute
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No